CLINICAL TRIAL: NCT05518071
Title: Intraoperative Near-infrared Fluorescence Imaging in Pancreatic- and Extrahepatic Bile Duct Tumors Using cRGD-ZW800-1 and Dedicated Imaging Systems: A Phase II Feasibility Testing, Dose-ranging and Optimal Dose-(Interval) Selection Trial
Brief Title: FLUOPANC-trial - Fluorescence-guided Surgery of Pancreatic and Bileduct Tumors Using cRGD-ZW800-1
Acronym: FLUOPANC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, dr. A.L. Vahrmeijer, MD, PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P21.128; 2019-004217-14 (EudraCT Number); NL 71219.058.22 (Other: Toetsingonline)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Adenocarcinoma; Cholangiocarcinoma
Keywords: Fluorescence Guided Surgery; Pancreatic Ductal Adenocarcinoma; Extrahepatic cholangiocarcinoma; Near-Infrared (NIR) Fluorescence imaging; Novel fluorescent probe; cRGD-ZW800-1
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Cohort 1 - N=4 (0.05mg/kg, 2-4h before intervention) (Experimental)
  Interventions: Drug: CRGD-ZW800-1; Device: Intraoperative near-infrared fluorescence imaging
- Cohort 2 - N=4 (0.05mg/kg, 14-24h before intervention) (Experimental)
  Interventions: Drug: CRGD-ZW800-1; Device: Intraoperative near-infrared fluorescence imaging
- Cohort 3 - N=4 (0.025mg/kg, 2-4h before intervention) (Experimental)
  Interventions: Drug: CRGD-ZW800-1; Device: Intraoperative near-infrared fluorescence imaging
- Cohort 4 - N=4 (0.025mg/kg, 14-24h before intervention) (Experimental)
  Interventions: Drug: CRGD-ZW800-1; Device: Intraoperative near-infrared fluorescence imaging
- Expansion cohort - N=4 (optimal dose, optimal dose-interval) (Experimental)
  Interventions: Drug: CRGD-ZW800-1; Device: Intraoperative near-infrared fluorescence imaging

INTERVENTIONS:
Drug: CRGD-ZW800-1 — Intravenous single bolus injection of the targeted NIR fluorophore cRGD-ZW800-1. This targeted 800nm zwitterionic fluorophore developed by the Hospital Pharmacy Department of LUMC consists of the fluorophore ZW800-1 conjugated to the cRGD peptide
Device: Intraoperative near-infrared fluorescence imaging — Intraoperative imaging will be performed with at least one of the following CE-marked near-infrared (NIR) fluorescence imaging systems: Quest Spectrum imaging platform (v2/3.0) for open-procedures, the Olympus or Karl-Storz system for the diagnostic laparoscopy or the Intuitive Surgical Da Vinci Xi (Firefly-mode) for minimally invasive robot-assisted procedures. With a NIR-imaging system a potential fluorescent signal of the tumor can be evaluated. Furthermore, the Quest Spectrum platform will also be used for evaluation of ex-vivo fluorescence of resected tissue on the back table (Back table imaging) and pathology department (ex-vivo imaging), which shall be performed during and after every procedure.

SUMMARY:
Pancreas as well as Cholangiocarcinoma have a dismal prognosis at time of diagnosis, due to late onset of clinical symptoms, patients present with advance disease. Complete surgical resection is the only potential curative treatment, however only a small percentage is eligible for upfront total surgical resection due to extension into anatomical related important vascular structures. Neoadjuvant chemo(radio)therapy has become the standard treatment modality for non-primary resectable disease (borderline resectable and locally advanced pancreatic cancer (LAPC)), where subsequent downstaging can make identification of the primary tumor more challenging during surgery. Near-infrared (NIR) fluorescence imaging can aid surgeons by providing real-time visualization of tumors, suspect lymph nodes and vital structures during surgery. Additional intra-operative feedback could possibly reduce the frequency of positive resection margins and increase complete removal of locally spread tumor and involved lymph nodes and could thereby improve patient outcomes as well as overall survival. cRGD-ZW800-1 is a targeted NIR-fluorophore, with specific binding capacity for integrins (αvβ3, αvβ5, αvβ6) which are overexpressed on tumor cells and tumor-associated vascular endothelium associated with neoangiogenesis.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most common causes of death in the United States. With a median survival of less than 6 months, the prognosis is very poor. After diagnosis, the 1 and 5-year survival rates are around 25% and 10%, respectively. Surgical resection is the only curative treatment, but also results in relatively low survival and present recurrence risk, depending on the stage. In the same order of magnitude, bile duct cancer is also found, it can be classified according to location within or outside the liver, extrahepatic bile duct tumors are much anatomically related to pancreatic tumors, surgical treatment is therefore often the same: (partial) pancreatic resection. During surgery, it is difficult to distinguish between malignant and benign tissue, especially if patients have been treated neoadjuvantly. Currently, near-infrared fluorescence imaging is a technique with great potential to illuminate important structures during surgery. Fluorescent substances can be injected intravenously, which then specifically attach to malignant cells or tumor-associated structures, such as stroma or blood vessels, and emit light in the near-infrared spectrum (700-900 nm). Thus, with specially equipped camera systems, tumors literally light up and the surgeon can completely remove the tumors during surgery in real time. cRGD-ZW800-1 is a newly developed fluorescent agent, which binds to integrins, which are associated with neoangiogenesis, and has the potential to make tumor cells in the pancreas more visible during surgery in order to achieve more complete surgical (R0) resections.

Aims of the study:

* To assess the feasibility, safety and tolerability of cRGD-ZW800-1 for the visualization of pancreatic carcinomas, perihilar or distal cholangiocarcinomas and if present associated metastatic lymph nodes and their distant metastases in real-time using specific NIR fluorescence imaging systems.
* Determining the optimal dose and dose interval of a single intravenous bolus injection of cRGD-ZW800-1 for intraoperative NIR imaging

Study design:

Open label, dose-ranging and optimal dose-(interval) selection study, with a two-factorial design. In total 20 patients diagnosed with a malignant tumor of the pancreas, or distal/hilar bile ducts, which are eligible for surgical resection with or without neoadjuvant treatment will be enrolled. These patients will be distributed over four dosing-, and one expansion cohort: Cohort 1 (0.05mg/kg, 2-4h before intervention), Cohort 2 (0.05mg/kg, 14-24h before intervention), Cohort 3 (0.025mg/kg, 2-4h before intervention), Cohort 4 (0.025mg/kg, 14-24h before intervention) and Cohort 5 (expansion cohort). Patients are included if they met the inclusion/exclusion criteria and will be screened during pre-operative work-up for surgery.

Study population: Patients with or without neoadjuvant treatment eligible for surgical resection at the Leiden University Medical Center (LUMC) of histologically proven malignant tumors of the pancreas head, neck and tail. As well as patients with histologically proven tumors of the peri-hilar and distal bile ducts (extrahepatic cholangiocarcinomas) with or without neoadjuvant treatment.

Intervention: Single bolus injection of cRGD-ZW800-1 2-24h before surgery. Intra-operative in-vivo assessment of NIR-fluorescence of tumor, lymph nodes, possible distant metastasis and anatomical related structures. After resection ex-vivo assessment of NIR-fluorescence of all resected tissue, on gross-macroscopy, bread loafs and microscopic slides.

Investigational drug: Intravenous single bolus injection of the targeted NIR fluorophore cRGD-ZW800-1. This targeted 800nm zwitterionic fluorophore developed by the Hospital Pharmacy Department of LUMC consists of the fluorophore ZW800-1 conjugated to the cRGD peptide.

Imaging: Intraoperative imaging will be performed with at least one of the following CE-marked near-infrared (NIR) fluorescence imaging systems: Quest Spectrum imaging platform (v2/3.0) for open-procedures, the Olympus or Karl-Storz system for the diagnostic laparoscopy or the Intuitive Surgical Da Vinci Xi (Firefly-mode) for minimally invasive robot-assisted procedures. With a NIR-imaging system a potential fluorescent signal of the tumor can be evaluated. Furthermore, the Quest Spectrum platform will also be used for evaluation of ex-vivo fluorescence of resected tissue on the back table (Back table imaging) and pathology department (ex-vivo imaging), which shall be performed during and after every procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old;
* Patients scheduled and eligible for open/robotic resection because of (histologically proven) pancreatic carcinoma with or without neoadjuvant treatment. As well as patients scheduled and eligible for resection because of (histologically proven) distal or perihilar cholangiocarcinoma with or without neoadjuvant treatment.
* All women of childbearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception for at least 30 days after their last dose of study treatment.
* Patients should be capable and willing to give informed consent before study specific procedures;

Exclusion Criteria:

* History of a clinically significant allergy or anaphylactic reactions;
* Patients with renal insufficiency (eGFR<60 ml/min/1,73 m2);
* Patients with a previous kidney transplantation in the medical history;
* Pregnant women, or women giving breast feeding;
* Patients who are immunocompromised and do not have the ability to respond normally to an infection due to an impaired or weakened immune system, caused by either a pre-existing disease or concomitant medications (excluding intended neoadjuvant treatment);
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Any condition that the investigator considers to be potentially jeopardizing the patients well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Visualization of the primary tumor using cRGD-ZW800-1 and dedicated NIR-Fluorescence imaging system. | Surgery
  Visualization is measured using the tumor-to-background ratio (TBR) in in-vivo and ex-vivo setting. A tumor-to-background ratio (TBR) of at least ≥1.5 provides sufficient contrast for adequate visualization/delineation and will therefore be used as cut-off value.

SECONDARY OUTCOMES:
Number and grade of treatment-emergent (serious) adverse events ((S)AEs). | Enrollment - EOS
Concordance between clinical assessment, histopathologic examination and NIR-Fluorescence imaging assessment of the resected tumor, lymph nodes and/or metastatic lesions and their histopathologic result. | Surgery
Define the optimal dose and dose interval of a single intravenous bolus injection of cRGD-ZW800-1. | Enrollment - EOS
  The optimal dose and ideal time window between administration of the study drug and intra-operative imaging during surgery will be assessed after all consecutive patients have been included, the endpoint for the combination of optimal dose and dose-interval is a tumor-to-background ratio of at least ≥1.5.
Tumor positive margins detected with NIR fluorescence imaging using cRGD-ZW800-1, referenced to histopathology. | Surgery
Number of tumor-positive lymph nodes and metastases detected by NIR fluorescence imaging using cRGD-ZW800-1, referenced to histopathology. | Surgery

OTHER OUTCOMES:
Exploratory endpoint | Surgery
  Fluorescence of fibrosis/tumor adjacent to the portal-venous structures (Superior Mesenteric Vein, Portal Vein) as well as the arterial structures (Communal Hepatic Artery, Celiac Trunk, Superior Mesenteric Artery) in patients who have received neoadjuvant chemotherapy for portal or arterial involvement (on previous scans).

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Valk KS, Deken MM, Handgraaf HJM, Bhairosingh SS, Bijlstra OD, van Esdonk MJ, Terwisscha van Scheltinga AGT, Valentijn ARPM, March TL, Vuijk J, Peeters KCMJ, Holman FA, Hilling DE, Mieog JSD, Frangioni JV, Burggraaf J, Vahrmeijer AL. First-in-Human Assessment of cRGD-ZW800-1, a Zwitterionic, Integrin-Targeted, Near-Infrared Fluorescent Peptide in Colon Carcinoma. Clin Cancer Res. 2020 Aug 1;26(15):3990-3998. doi: 10.1158/1078-0432.CCR-19-4156. Epub 2020 Apr 28. PMID 32345649
- [Background] Handgraaf HJM, Boonstra MC, Prevoo HAJM, Kuil J, Bordo MW, Boogerd LSF, Sibinga Mulder BG, Sier CFM, Vinkenburg-van Slooten ML, Valentijn ARPM, Burggraaf J, van de Velde CJH, Frangioni JV, Vahrmeijer AL. Real-time near-infrared fluorescence imaging using cRGD-ZW800-1 for intraoperative visualization of multiple cancer types. Oncotarget. 2017 Mar 28;8(13):21054-21066. doi: 10.18632/oncotarget.15486. PMID 28416744